CLINICAL TRIAL: NCT01054508
Title: Effect of Tredaptive on Serum Lipoproteins, Lipoproteins Metabolism, Oxidative Stress and HDL Antioxidant Function
Brief Title: Effect of Tredaptive on Serum Lipoproteins and Inflammatory Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRED012010; R01049 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Placebo (4 weeks) --> Placebo (12 weeks) --> Placebo (4 weeks) --> Tredaptive (12 weeks) (Other): Placebo (4 weeks) --> Placebo (12 weeks) --> Placebo (4 weeks) --> Tredaptive (12 weeks) There were two interventional periods of 12 weeks during which patients received either Placebo or Tredaptive (nicotinic acid/laropiprant). Patient who received Tredaptive were given dosages of 1g/20mg for 4 weeks followed by 2g/40mg for 8 weeks.
  Interventions: Drug: nicotinic acid/laropiprant
- Arm 2: Placebo (4 weeks) --> Tredaptive (12 weeks) --> Placebo (4 weeks) --> Placebo (12 weeks) (Other): Placebo (4 weeks) --> Tredaptive (12 weeks) --> Placebo (4 weeks) --> Placebo (12 weeks) There were two interventional periods of 12 weeks during which patients received either Placebo or Tredaptive (nicotinic acid/laropiprant). Patient who received Tredaptive were given dosages of 1g/20mg for 4 weeks followed by 2g/40mg for 8 weeks.
  Interventions: Drug: nicotinic acid/laropiprant

INTERVENTIONS:
Drug: nicotinic acid/laropiprant — Nicotinic acid/laropiprant (1g/20mg) daily for 4 weeks, then nicotinic acid/laropiprant (2g/40mg) daily for 8 weeks.
  Other Names: Tredaptive

SUMMARY:
Cardiovascular disease (CVD) is associated with high levels of low-density lipoprotein (LDL) cholesterol and low levels of high-density lipoprotein (HDL) cholesterol.

CVD results from 'hardening of the arteries' when there is a build-up of cholesterol in the walls of blood vessels. LDL is the main carrier of cholesterol in the body. LDL particles are responsible for transporting cholesterol that is deposited in vessel walls. LDL particles can also be altered in structure and turn into an irritant to the vessel walls. The body responds to the irritating effect of LDL by producing substances that result in inflammation. This sequence of events eventually leads to the vessels becoming permanently damaged. HDL has a protective role in CVD. It is associated with the enzyme paraoxonase which protects the body from the damaging effects of altered LDL particles.

Nicotinic acid (niacin) has the ability to lower LDL levels and raise HDL levels thus reducing the incidence of CVD. Our study aims to show that niacin not only has good effects on cholesterol levels but is also able to reduce inflammation. Niacin is often poorly tolerated due to flushing side effect. Tredaptive is a formulation that combines niacin with laropiprant, an agent that reduces flushing hence improving tolerability and compliance.

Patients who are receiving cholesterol-lowering medication and whose LDL levels have not reached the recommended target are recruited to the study. The study will be conducted at the Manchester Royal Infirmary. The study has two consecutive 16 week periods. In each period patients will be randomised to either tredaptive or placebo. They will attend for 5 monitoring visits. Apart from the first visit, fasting blood samples will be taken from them during all subsequent visits.

DETAILED DESCRIPTION:
The design is a placebo-controlled cross-over study. The study has 2 consecutive 16 week periods. If a patient satisfies the inclusion/exclusion criteria and consents to participate in the study, he/she will enter a 4-week placebo run-in period. This is followed by a 12-week treatment period where the patient will be assigned tredaptive or placebo randomly. At the end of the treatment period the patient will enter a second 4-week placebo period before going onto the second 12-week treatment period. Patients who are randomised to placebo in the first treatment period will receive tredaptive in the second treatment period and vice versa. Thus all participating patients will receive active medication for one treatment period in the study.

Patients will continue taking statins for the duration of the study, ensuring the cholesterol-lowering benefits they have from their usual medication are not compromised.

Patients will be recruited from the Lipid Clinic at the Manchester Royal Infirmary. The study will be explained fully to the patients who will have time to ask questions. Information leaflets will be given to patients who will be encouraged to take at least 1 day to discuss the study with their families, friends and general practitioners before consenting.

The study comprises 5 visits. At the first visit, informed consent will be taken from the patients. The visit also includes history taking and physical examination. Subsequent visits take place at the end of 4th and 16th weeks. This is repeated for the second 16 week period. Apart from the first visit, patients will be required to give a blood sample of 50 ml at each of the visits. They will be asked to fast overnight (from 22.00 hours) the day before the visit and blood sampling will be done before midday the following day. Blood will be taken by an experienced doctor or nurse and the only risks involved may be bruising at the puncture site.

ELIGIBILITY:
Inclusion Criteria:

-Men and women who are taking cholesterol-lowering medication (maximum tolerated statins and/or ezetimibe) and who have not reached the recommended LDL target of less than 1.8 mmol/l (70 mg/l). Ezetimibe will be stopped 4 weeks before entering the study.

Exclusion Criteria:

* Pregnant and/or breast-feeding women.
* Significant renal impairment (eGFR < 59ml/min).
* Active liver disease and transaminases > 3 times upper limit of normal range.
* Patients on fibrates.
* Patients on Omacor.
* Patients who are allergic to nicotinic acid.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in HDL Levels | 14 months
  As exactly listed in the protocol, the primary outcome will be changes in HDL-C level. The mean value will be assessed before and after treatment. This level will be compared to the mean value between the placebo and Tredaptive groups.

SECONDARY OUTCOMES:
Changes in paraoxonase activity | 14 months
  Changes in PON1
Changes in LDL | 14 months
  Changes in oxidised LDL and glycated LDL
Changes in HDL inflammatory index | 14 months
  Changes in HDL inflammatory index

CONTACTS AND LOCATIONS:
Overall Officials: Handrean Soran, MRCP, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom

REFERENCES:
- [Derived] Yadav R, Liu Y, Kwok S, Hama S, France M, Eatough R, Pemberton P, Schofield J, Siahmansur TJ, Malik R, Ammori BA, Issa B, Younis N, Donn R, Stevens A, Durrington P, Soran H. Effect of Extended-Release Niacin on High-Density Lipoprotein (HDL) Functionality, Lipoprotein Metabolism, and Mediators of Vascular Inflammation in Statin-Treated Patients. J Am Heart Assoc. 2015 Sep 15;4(9):e001508. doi: 10.1161/JAHA.114.001508. PMID 26374297